CLINICAL TRIAL: NCT01973543
Title: An Open-label Safety and Efficacy Study of VY-AADC01 Administered by MRI-Guided Convective Infusion Into the Putamen of Subjects With Parkinson's Disease With Fluctuating Responses to Levodopa
Brief Title: Safety Study of AADC Gene Therapy (VY-AADC01) for Parkinson's Disease
Acronym: AADC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: University of California, San Francisco (Other); Veristat, Inc. (Other); Feinstein Institute for Medical Research (Other); Oregon Health and Science University (Other); Voyager Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PD-1101; 1302-1209 (Registry Identifier: NIH OBA)
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Parkinson's Disease
Keywords: PD; Parkinson's disease; Aromatic Amino Acid Decarboxylase; AADC; AAV2-AADC; AAV2; Viral Vector; Gene Therapy; Gene Transfer; MRI; PET; VY-AADC01
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: VY-AADC01
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VY-AADC01 Dose 1 (Experimental): 7.5 x 10^11 vector genomes of VY-AADC01; Single dose, neurosurgically infused, bilaterally into the striatum.
  Interventions: Biological: VY-AADC01
- VY-AADC01 Dose 2 (Experimental): 1.5 x 10^12 vector genomes of VY-AADC01; Single dose, neurosurgically infused, bilaterally into the striatum.
  Interventions: Biological: VY-AADC01
- VY-AADC01 Dose 3 (Experimental): 4.7x 10^12 vector genomes of VY-AADC01; Single dose, neurosurgically infused, bilaterally into the striatum.
  Interventions: Biological: VY-AADC01

INTERVENTIONS:
Biological: VY-AADC01 — Neurosurgical delivery of VY-AADC01 to the brain.
  Other Names: AAV2-hAADC

SUMMARY:
Safety study of AADC gene transfer (VY-AADC01) in subjects with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease is a neurodegenerative disorder involving loss of neurons that release dopamine in the striatum. To compensate for the loss of dopamine, patients are typically prescribed levodopa medication which is converted to dopamine by the enzyme Aromatic L-Amino Acid Decarboxylase (AADC). As Parkinson's disease progresses, levodopa therapy becomes less effective and is associated with motor fluctuations, involuntary movements and other complications.

This study will primarily investigate the safety of increasing AADC levels in the striatum via AADC gene delivery. The hAADC gene is packaged into a gene transfer vector derived from a common, non-pathogenic virus (AAV2) to which >90% of humans have been exposed. This investigational drug, termed VY-AADC01, will be injected directly into the striatum during a neurosurgical procedure that is performed with real-time MRI imaging to monitor delivery.

Subjects will continue to take Parkinson's disease medications, including levodopa.

The safety and potential clinical responses to VY-AADC01 will be assessed by repeated clinical evaluations of Parkinson's disease, cognitive tests, laboratory blood tests and neuroimaging. Clinical evaluations will be performed over a 3 year follow-up period. A test to specifically assess the clinical response to levodopa will be performed once before AADC gene delivery and approximately 6 months after.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's disease
* Disease duration of at least 5 years or more
* Adequate duration of levodopa therapy
* Modified Hoehn and Yahr Staging of at least 2.5 in the OFF state
* Candidate for surgical intervention because of disabling motor complications.
* UPDRS Part III (total motor) score ≥ 25 and a maximum of 60 in the OFF state.
* Unequivocal responsiveness to dopaminergic therapy.
* Stable Parkinson's symptoms and medication regimen for at least 4 weeks prior to screening examination.
* Ability to comprehend and sign the informed consent.
* Normal Laboratory values prior to surgery.
* Neutralizing AAV2 antibody titer ≤ 1:1200
* Ability to travel to study visits alone or able to designate a caregiver.
* Subject agrees to defer any neurological surgery, including deep brain stimulation, until after completing the 12 month study visit (unless recommended by study neurologist).
* Subject agrees to not participate in any other therapeutic intervention study for 12 months after surgery.
* Subject agrees to not have any vaccinations within 30 days of surgery.

Exclusion Criteria:

* Atypical or secondary parkinsonism, including but not limited to symptoms believed to be due to trauma, brain tumor, infection, cerebrovascular disease, other neurological disease, or to drugs, chemicals or toxins.
* Presence of dementia as defined by a Mattis Dementia Rating Scale-Second Edition (MDRS-2) of less than 130 at screening.
* Presence or history of psychosis, with the exception of mild, benign hallucinations believed in the judgment of the investigators to be related to Parkinson's medications.
* Presence of severe depression as measured by Beck Depression Inventory II (BDI-II) > 28 or a history of a major affective disorder within 5 years of screening examination.
* Current suicidal ideation or suicide attempt within 5 years of screening examination.
* History of substance abuse within 2 years of screening examination.
* Brain imaging abnormalities in the striatum or other regions that would substantially increase risk of surgery.
* Contraindication to MRI and/or gadoteridol.
* Coagulopathy or inability to temporarily stop any anticoagulation or antiplatelet prior to surgery.
* Prior brain surgery including deep brain stimulation, infusion therapies or any other brain surgery.
* Prior gene transfer.
* History of stroke, poorly controlled or significant cardiovascular disease, diabetes or any other acute or chronic medical condition.
* History of malignancy other than treated carcinoma in situ within three years of screening evaluation.
* Clinically apparent or laboratory-detected infection.
* Prior or current treatment with any investigational agent within 2 months of screening evaluation.
* Chronic immunosuppressive therapy, including chronic steroids, immunotherapy, cytotoxic therapy and chemotherapy.
* Pregnant and lactating women.
* Subject with reproductive capacity who is unwilling to use barrier contraception.
* Any medical condition that is likely to lead to disability during the course of the study and interfere with confound study assessments
* Any factors, medical, or social, which would likely cause the subject to be unable to follow the study protocol, including geographical inaccessibility.
* Ongoing treatments such as, neuroleptic medications, apomorphine, or levodopa infusion therapy (Duodopa®).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Safety of AADC Gene Transfer | 3 Years after Gene Transfer
  Safety and Tolerability of AADC Gene Transfer assessed by Adverse Events and Serious Adverse Events.

SECONDARY OUTCOMES:
Parkinson's Symptoms | 3 Years after Gene Transfer
  Effect of AAV2-hAADC on Parkinson's symptoms as recorded in subject diaries, neurological, motor, and non-motor assessments, quality of life surveys and changes to Parkinson's medications.
PET Scan Imaging | 6 Months after Gene Transfer
  Relationship between AAV2 distribution in the brain and change in AADC expression as seen in PET imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Hersch, MD, Study Director — Voyager Therapeutics
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christine CW, Richardson RM, Van Laar AD, Thompson ME, Fine EM, Khwaja OS, Li C, Liang GS, Meier A, Roberts EW, Pfau ML, Rodman JR, Bankiewicz KS, Larson PS. Safety of AADC Gene Therapy for Moderately Advanced Parkinson Disease: Three-Year Outcomes From the PD-1101 Trial. Neurology. 2022 Jan 4;98(1):e40-e50. doi: 10.1212/WNL.0000000000012952. Epub 2021 Oct 14. PMID 34649873
- [Derived] Christine CW, Bankiewicz KS, Van Laar AD, Richardson RM, Ravina B, Kells AP, Boot B, Martin AJ, Nutt J, Thompson ME, Larson PS. Magnetic resonance imaging-guided phase 1 trial of putaminal AADC gene therapy for Parkinson's disease. Ann Neurol. 2019 May;85(5):704-714. doi: 10.1002/ana.25450. Epub 2019 Mar 26. PMID 30802998
- See also: Voyager website — http://www.voyagertherapeutics.com